CLINICAL TRIAL: NCT04303715
Title: No Axillary sUrgical Treatment In Clinically Lymph Node Negative Patients After UltraSonography[NAUTILUS]: A Prospective, Multicenter, Phase III Clinical Trial
Brief Title: No Axillary sUrgical Treatment In Clinically Lymph Node Negative Patients After UltraSonography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAUTILUS study
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No SLNB group (Experimental): The study arm - BCS without SLNB
  Interventions: Procedure: No SLNB
- SLNB group (Other): The Control Arm - BCS with SLNB(+/-ALND)
  Interventions: Procedure: SLNB

INTERVENTIONS:
Procedure: No SLNB — BCS only. Ommission of SLNB by axilla ultrasonography among selective breast cancer patients
  Arms: No SLNB group
Procedure: SLNB — BCS with SLNB(+/-ALND)
  Arms: SLNB group

SUMMARY:
NAUTILUS study is a prospective, multicenter, RCT. Clinically T1,T2, node negative BCS candidates with no evidence of metastases in AUS are 1:1 randomized into no SLNB group and SLNB group.

NAUTILUS study aim to establish the minimally invasive treatment of breast cancer by reexamining the necessity of sentinel lymph node biopsy among patients with invasive breast cancer who have tumors under 5cm, are clinically node-negative, and are having breast conserving surgery performed.

DETAILED DESCRIPTION:
[Background] Skipping ALND, the follow-up treatment in SN-positive patients, has non-inferior oncological outcomes compared to SLNB-only group, given that there is no severe SN metastases.

Axillary ultrasound can effectively exclude high nodal burden, showing 95% NPV in a systematic review.

SLNB has morbidity including lymphedema, limited range of motion, pain, and other post-surgical complications, eventually leading to reduced quality of life.

Considering improvement of imaging modalities and adjuvant care, survival outcome of SLNB must be re-evaluated. Especially research reflective of the regional specificities of Korea and Asia-Pacific is needed.

[Study design] Prospective, Multicenter, RCT.

[Statistical considerations] According to Z0011 trial, 5yr DFS in eligible patients is expected to be 86%, which is between previous data of 88.6% in cT1,2 and SN-negative patients4, and 83.9% in cT1,2 and 1-2 SN-positive patients.

Non-inferiority margin is set at 5%. With 5% significance level and 80% power, 780 patients are needed in each group. Assuming a 10% drop out rate, 1734 patients need to be recruited.

[Screening and Randomization] Participants undergo screening tests that assess eligibility according to inclusion/exclusion criteria.

In order to identify axillary lymph node metastases, axillary ultrasound is first performed by radiologists. Patients showing normal features are enrolled, while for conditionally normal patients, with only 1 suspicion of low nodal burden, axillary lymph node biopsy should be performed. Suspicious patients are excluded under following conditions: patients with 1 or more suspicion of high nodal burden, 2 or more suspicion of low nodal burden, or T2 invasive lobular carcinoma patients with 1 or more low nodal burden. The severity of nodal burden is defined through the criteria.

Patients who underwent radiological axillary staging are randomly assigned (1:1) to the study arm and the control arm before surgical care. Stratification is done based on trial centers and tumor sizes.

[Post-surgical care] All patients are planned to receive ipsilateral whole breast radiation. Patients randomized to non-SLNB arm are recommended to follow high tangential radiotherapy protocol, in which upper margin of radiation field includes axillary level I and II or lies within 2CM from humeral head.

Additional treatment may be performed if deemed necessary by the researcher

[Objectives]

1. Primary objective

   - 5yr invasive Disease Free Survival
2. Secondary objectives

   * 5yr Overall Survival
   * 5yr Distant Metastasis Free Survival
   * Axillary recurrence rate
   * Patient reported AE
   * QoL

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 19 years
* Invasive unilateral breast carcinoma with histological confirmation
* History of invasive breast cancer
* Histologically or radiologically no suspicion of distant metastases
* Performance status corresponding to ECOG grade 0-2
* Tumor size clinically and radiologically ≤ 5cm, independent of hormone receptor and HER2 status
* Clinically and sonographically negative axillary lymph nodes before biopsy; core needle biopsy or fine needle aspiration of suspicious lymph node required
* BCS candidate with postoperative whole-breast irradiation and adequate systemic therapy
* No psychological and geographical restriction in follow-up
* Written informed consent

Exclusion Criteria:

* History of any cancer in the previous 5 years
* Bilateral breast cancer
* Invasive breast cancer treated with neoadjuvant therapy
* Tumor size clinically and radiologically > 5cm
* Mastectomy candidate
* Pregnancy and breastfeeding
* Male breast cancer
* Unable to understand and fill out questionnaires

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1734 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
invasive Disease Free Survival (iDFS) | 5 years
  Evaluate invasive disease free survivals

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Evaluate overall survival
Distant Metastasis Free Survival (DMFS) | 5 years
  Evaluate distant metastasis free survival
Axillary recurrence rate | 5 years
  Evaluate ipsilateral axillary recurrence rate
Locoregional Recurrence Rate (LRR) | 5 years
  Evaluate locoregional recurrence rate
Patient reported Adverse Events (AEs) | 1 year
  Evaluate Patient reported Adverse Events
QoL | 1 year
  Evaluate Quality of Life of patient by EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jung JG, Ahn SH, Lee S, Kim EK, Ryu JM, Park S, Lim W, Jung YS, Chung IY, Jeong J, Chang JH, Shin KH, Chang JM, Moon WK, Han W. No axillary surgical treatment for lymph node-negative patients after ultra-sonography [NAUTILUS]: protocol of a prospective randomized clinical trial. BMC Cancer. 2022 Feb 20;22(1):189. doi: 10.1186/s12885-022-09273-1. PMID 35184724
- [Derived] Chang JM, Shin HJ, Choi JS, Shin SU, Choi BH, Kim MJ, Yoon JH, Chung J, Kim TH, Han BK, Kim HH, Moon WK. Imaging Protocol and Criteria for Evaluation of Axillary Lymph Nodes in the NAUTILUS Trial. J Breast Cancer. 2021 Dec;24(6):554-560. doi: 10.4048/jbc.2021.24.e47. Epub 2021 Nov 24. PMID 34877830